CLINICAL TRIAL: NCT01742962
Title: Prevalence of Neglected Side Effects to Radical Prostatectomy
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-58-0015 / HEH.750.19-31; H-2-2012-FSP43 (Other: Denmark: The Regional Committee on Biomedical Research Ethics)
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Prostate Cancer
Keywords: Prostatectomy; Prostate cancer; Orgasm; Urinary incontinence; Climacturia(orgasm related urinary incontinence); Penis; Dysorgasmia (pain in relation to orgasm); Pain; Anorgasmia; Penile shortening; Erectile dysfunction
MeSH Terms: conditions — Prostatic Neoplasms; Orgasm; Urinary Incontinence; Pain; Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radical prostatectomy for prostate cancer: Prior treatment with open or robot assisted laparoscopic prostatectomy.
  Interventions: Procedure: Radical prostatectomy for prostate cancer

INTERVENTIONS:
Procedure: Radical prostatectomy for prostate cancer — Prior treatment with open or robot assisted laparoscopic prostatectomy.

SUMMARY:
The purpose of this exploratory data collection is to strengthen our knowledge of some of the rarer distresses following surgical removal of the prostate. In general these are:

* Side effects related to sexuality, including:
* Altered perception of orgasm,
* Orgasm associated pain,
* Penile shortening and deformity.
* Side effects related to urinary incontinence.
* Urinary tract infection after operation.
* Influence of distress on sexual quality of life.
* Influence of distress on the patient´s sex drive.

In addition information on a range of demographics and information on the patient´s erectile function will be collected.

DETAILED DESCRIPTION:
Approximately 1 out of 6 men will, at some point of their life become diagnosed with prostate cancer. Treatment options included medication therapy, radiation therapy, and surgery. This data collection aims to gather information on some of the lesser known distresses experienced by patients following surgical removal of the prostate gland.

Erectile dysfunction and urinary incontinence remain common, but thoroughly investigated side effects. Thus they will not be of primary interest here, but considered factors for correlation. During the last couple of years, a series of lesser known side effects have come to investigators attention. These include altered perception of orgasm, orgasm related pain, sexual-related urinary incontinence, and shortening -and impairing deviations of the penis. Few studies have investigated these side effects, and clear knowledge of why, and how often these problems arise, remain scarce. This study will contribute to that knowledge.

In addition, the questionnaire will include a series of exploratory questions, concerning lower urinary tract infections, treatment satisfaction, alcohol and urinary incontinence, reasons for abandoning treatment for erectile dysfunction, and an assessment of libido prior to and after radical prostatectomy.

The data collection will include approximately 400 patients from the department of urology at the University Hospital in Herlev, Copenhagen, Denmark. A questionnaire will be sent to patients together with a stamped addressed envelope in order to optimize the response rate. Results will be kept in a separate database from personal information.

ELIGIBILITY:
Inclusion Criteria:

* All patient who have undergone radical prostatectomy at the department of urology, Copenhagen University Hospital, Herlev, between 3 months and 3 years before initiation of the study.

Exclusion Criteria:

* Incontinence associated with sexual activity Prior to surgery
* Peyronies disease Prior to surgery
* Orgasm related pain Prior to surgery
* Anorgasmia Prior to surgery

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Post prostatectomy patients operated at Copenhagen University Hospital in Herlev, Denmark.
Sampling Method: Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Urinary incontinence in relation to sexual activity measured as percentage of the population. | A momentary exploratory analysis of the problem in the study population, who are between 3 months and 3 years post radical prostatectomy.
  The percentage of the study population experiencing urinary incontinence when engaging in sexual activity.
Incidence of altered perception of orgasm measured as percentage of the population. | A momentary exploratory analysis of the problem in the study population, who are between 3 months and 3 years post radical prostatectomy.
  The percentage of the study population experiencing altered perception of orgasm.
Incidence of orgasm related pain measured as percentage of the population. | A momentary exploratory analysis of the problem in the study population, who are between 3 months and 3 years post radical prostatectomy.
  The percentage of the study population experiencing orgasm related pain.
Incidence of impairing deviations or loss of length of the penis measured as percentage of the population. | A momentary exploratory analysis of the problem in the study population, who are between 3 months and 3 years post radical prostatectomy.
  The percentage of the study population experiencing impairing deviations or loss of length of the penis.

OTHER OUTCOMES:
Incidence of lower urinary tract infections following radical prostatectomy | A momentary exploratory analysis of the problem in the study population, who are between 3 months and 3 years post radical prostatectomy.
  We want to know how large a percentage of patients treated with radical prostatectomy are experiencing a lower urinary tract infection post surgery.
Incidence of alcohol related incontinence in patients undergone radical prostatectomy | A momentary exploratory analysis of the problem in the study population, who are between 3 months and 3 years post radical prostatectomy.
  Does alcohol exacerbate incontinence symptoms?
Impact of radical prostatectomy on the patients libido. | A momentary exploratory analysis of the problem in the study population, who are between 3 months and 3 years post radical prostatectomy.
  Does radical prostatectomy influence patients libido?
Patterns of use and discontinuation of use of aids for erectile dysfunction. | A momentary exploratory analysis of the problem in the study population, who are between 3 months and 3 years post radical prostatectomy.
  A series of questions will investigate the patients use of aids for erectile dysfunction and reasons for discontinuation.
Patient satisfaction with treatment. | A momentary exploratory analysis of the problem in the study population, who are between 3 months and 3 years post radical prostatectomy.
  Assessed by a global satisfaction scale, and an evaluation of fulfillment of expectations prior to treatment.
How do the patients gather knowledge of their disease? | A momentary exploratory analysis of the problem in the study population, who are between 3 months and 3 years post radical prostatectomy.
  From which sources do the patients get their knowledge of prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Anders U. K. Frey, Stud.Med., Principal Investigator — Copenhagen University Hospital in Herlev, Denmark; Mikkel M. Fode, Dr., Study Director — Copenhagen University Hospital in Herlev, Denmark; Jens Sønksen, Professor, Study Chair — Copenhagen University Hospital in Herlev, Denmark
Locations (1):
- Copenhagen University Hospital in Herlev, Denmark, Herlev, Herlev, Denmark